CLINICAL TRIAL: NCT04655690
Title: A Trial Investigation the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneous NNC0471-0119 in Subjects With Type 1 Diabetes Mellitus
Brief Title: A Study to Look at How Safe Insulin NNC0471-0119 is and How it Works in People With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1471-4612; U1111-1247-7440 (Other: World Health Organization (WHO)); 2020-000665-16 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2020-10-28; First posted 2020-12-07 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NNC0471-0119 (Experimental): Participants randomised to NNC0471-0119
  Interventions: Drug: NNC0471-0119
- Faster aspart (Active Comparator): Participants randomised to faster aspart.
  Interventions: Drug: Fast-acting insulin aspart

INTERVENTIONS:
Drug: NNC0471-0119 — Participants will be randomised to either of five dose levels 0.3, 0.6, 1.2, 2.4 or 3.6 of NNC0471-0119 nanomol per kilogram body weight, which will be administered as a single dose. NNC0471-0119 will be administered subcutaneously (s.c., under the skin) in fasting state.
  Arms: NNC0471-0119
Drug: Fast-acting insulin aspart — Participants will get a fixed dose of 0.2 units of fast-acting insulin aspart (Fiasp®) per kilogram body weight, administered subcutaneously (s.c., under the skin) in fasting state.
  Arms: Faster aspart

SUMMARY:
This study is looking at the safety of the new medicine, insulin NNC0471-0119, its concentrations in the blood and effect on blood sugar for the treatment of type 1 diabetes. Insulin NNC0471-0119 will be compared to faster aspart. The purpose of this study is to test how insulin NNC0471-0119 is tolerated by participants body, how it is transported in participants bloodstream, how long it stays there and how the blood sugar is lowered compared to faster aspart. Participants will get either the new insulin NNC0471-0119 or faster aspart-which treatment participants get is decided by chance. It is the first time insulin NNC0471-0119 is tested in people. Faster aspart is a globally used medication for treatment of diabetes mellitus. Participants will get one single injection in a fasting state which will take place at the study site. The medicine will be injected under the skin in the stomach. The study will last for about 13-53 days, depending on individual visit schedule. Participants will have four clinic visits with the study doctor, one of which will require an in-house visit period of 3 days. During the in-house visit, two intravenous cannulas will be inserted for sampling of blood and infusion of insulin. Participants cannot be in the study if the study doctor thinks that there are risks to their health. Women: Women cannot take part if they are of childbearing potential.

ELIGIBILITY:
Inclusion Criteria:

* Male subject or female subject of non-childbearing potential. Non-childbearing potential being defined as surgically sterilised (i.e. documented hysterectomy, bilateral salpingectomy or bilateral oophorectomy) or being postmenopausal (defined as no menses for 12 months without an alternative medical cause) prior to the day of screening.
* Aged 18-55 years (both inclusive) at the time of signing informed consent.
* Diagnosed with Type 1 Diabetes Mellitus (T1DM) greater than or equal to 1 year prior to the day of screening.
* Current total daily bolus insulin treatment less than 0.7(I)U/kg/day.

Exclusion Criteria:

* Known or suspected hypersensitivity to investigational medicinal products (IMPs) or related products.
* Participation in any clinical trial of an approved or non-approved IMP within 90 days before screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AEs) | From investigational medicinal product (IMP) administration at day 1 (Visit 2) and up to 22 days post IMP administration (Visit 3)
  Number of events

SECONDARY OUTCOMES:
Number of hypoglycaemic episodes | 0 to 24 hours after IMP administration
  Number of episodes
AUCNNC0471-0119,0-30 min/AUCNNC0471-0119,0-t: Ratio of the area under the serum NNC0471-0119 concentration-time curve from 0-30 min and 0-t, where t is the last observed time point with insulin concentration above lower limit of quantification (LLOQ). | 0 to 12 hours after IMP administration
  % (Percent)
AUCNNC0471-0119,2h-t/AUCNNC0471-0119,0-t: Ratio of the area under the serum NNC0471-0119 concentration-time curve from 2 hours to t and 0 to t, where t is the last observed time point with insulin concentration above LLOQ. | 0 to 12 hours after IMP administration
AUCNNC0471-0119, 0-t: Area under the serum NNC0471-0119 concentration-time curve from 0 to t, where t is the last observed time point with insulin concentration above LLOQ. | 0 to 12 hours after IMP administration
  h*pmol/L
Cmax,NNC0471-0119: Maximum observed serum NNC0471- 0119 concentration | 0 to 12 hours after IMP administration
  pmol/L
tmax,NNC0471-0119: Time to maximum observed serum NNC0471-0119 concentration | 0 to 12 hours after IMP administration
  Minutes
t½, NNC0471-0119: Terminal half-life for NNC0471-0119 | 0 to 12 hours after IMP administration
  Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com